CLINICAL TRIAL: NCT00507364
Title: Treatment of Anal Fissure by Activated Human Macrophages
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: qwerty-HMO-CTIL
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: Biological Therapy for Chronic Anal Fissure; Treatment by Biological Factors - Activated Macrophages; Interventional Study

INTERVENTIONS:
Drug: Local injection of activated macrophages to anal fissure

SUMMARY:
Chronic anal fissure is a linear tear in the distal anal canal. Most chronic fissures require intervention to heal. Surgical sphincterotomy is currently performed. However, the procedure permanently weakens the internal sphincter and may be associated with permanent complications such as incontinence. Current topical treatment or " chemical sphincterotomy" is effective in the short term for about 70% of the patient more than 50% of them will suffer from recurrence. Number of studies support the hypothesis that local ischemia is the reason for failure to heal in anal fissure. Treatment of refractory wounds by macrophage suspension is an innovative method since 1995, macrophage suspensions have been used successfully in more than 1400 patients in several hospitals in Israel without any side effect.Macrophages have key function in almost every stage of wound healing. They help in the digestion of bacteria, in a later stage, they secret IL-6, which influences endothelial cell proliferation and the initiation of angiogenesis.

The study hypothesis is that local injection of activated human macrophages into chronic anal fissure may induce fissure healing.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive symptomatic adults with chronic idiopathic anal fissure

Exclusion Criteria:

* Pregnant women
* Acute fissures
* Anal fissures of various causes ( i.e.,hemorrhoids, fistula in ano, inflammatory bowel disease)
* Immunosuppressed patients

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
COMPLETE FISSURE HEALING

CONTACTS AND LOCATIONS:
Overall Officials: Yosef (Joseph) Lysy, MD, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital Gastroenterology Unit, Jerusalem, Israel

REFERENCES:
- [Result] Danon D, Madjar J, Edinov E, Knyszynski A, Brill S, Diamantshtein L, Shinar E. Treatment of human ulcers by application of macrophages prepared from a blood unit. Exp Gerontol. 1997 Nov-Dec;32(6):633-41. doi: 10.1016/s0531-5565(97)00094-6. PMID 9785089